CLINICAL TRIAL: NCT07188337
Title: Examining the Demographic, Clinical, and Laboratory Data of Patients With Diabetic Foot Ulcers Admitted to 5 Azar Hospital in 2024 (Registry Project)
Brief Title: Characteristics of Diabetic Foot Ulcer Patients
Status: Recruiting | Type: Observational
Sponsor: Golestan University of Medical sciences (Other)
Responsible Party: Principal Investigator, Pezhman Kharazm, MD, Assistant Professor of Vascular Surgery, Golestan University of Medical Sciences, Golestan University of Medical sciences
Other Study IDs: 114627
Record Dates: First submitted 2025-08-31; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcer; Diabetes Complications
Keywords: diabetic foot ulcer; diabetes mellitus; amputation; neuropathy
MeSH Terms: conditions — Diabetic Foot; Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study examines the demographic, clinical, and laboratory characteristics of patients with diabetic foot ulcers admitted to 5 Azar Hospital, Gorgan, in 2024. By analyzing factors such as Hb, WBC, HbA1C, ESR, and CRP in relation to ulcer severity, the study aims to identify predictors of outcomes and support more effective prevention and management strategies

DETAILED DESCRIPTION:
Diabetic foot ulcer (DFU) is one of the most serious and preventable complications in diabetic patients, often leading to infection, hospitalization, lower limb amputation, and increased mortality. This cross-sectional descriptive-analytical study aims to investigate the demographic, clinical, and laboratory characteristics of approximately 200 patients with DFU admitted to 5 Azar Hospital, Gorgan, in 2024. Data will be retrospectively collected from medical records after obtaining ethical approval.

The study will analyze relationships between patient demographics, clinical features, and laboratory findings (including Hb, WBC, HbA1C, ESR, CRP) with ulcer severity based on Wagner's classification. Statistical tests such as independent t-test, chi-square, Fisher's exact test, and multivariable logistic regression will be used.

By identifying key factors associated with ulcer severity and outcomes, the findings of this study may contribute to more effective prevention and management strategies for diabetic foot ulcers, ultimately reducing complications and healthcare costs

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to 5 Azar Hospital, Gorgan, in 2024
* Diagnosis of diabetic foot ulcer (DFU) confirmed by medical records
* Complete demographic, clinical, and laboratory data available in medical files

Exclusion Criteria:

* Incomplete or missing medical records
* Patients with foot ulcers of non-diabetic etiology
* Patients whose key laboratory data are unavailable

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of approximately 200 patients with diabetic foot ulcers admitted to 5 Azar Hospital, Gorgan, during 2024. Patients will be identified retrospectively from hospital medical records. Both demographic and clinical data, as well as laboratory findings, will be extracted for analysis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Severity of diabetic foot ulcer (measured by Wagner classification at admission) | Baseline
  Measured by Wagner classification
Laboratory parameters and ulcer grade | Baseline
  Association between Hb, WBC, HbA1C, ESR, and CRP levels with Wagner ulcer grade

SECONDARY OUTCOMES:
Duration of diabetes until ulcer onset | Baseline
  Time (in years) between diabetes diagnosis and first DFU occurrence
Smoking status and ulcer severity | Baseline
  Correlation between smoking history (yes/no) and Wagner ulcer grade
Treatment outcomes | At hospital discharge (average of 10 days)
  Frequency of outcomes: antibiotic therapy, wound debridement, or amputation
Ulcer recurrence | During 12-month follow-up (based on records)
  Number of hospital readmissions due to DFU.
Demographic distribution | Baseline
  Age, sex, occupation, and ethnicity of DFU patients

CONTACTS AND LOCATIONS:
Locations (1):
- 5Th Azar Medical Center, Gorgan, Outside of the US, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol